CLINICAL TRIAL: NCT03353181
Title: Application of Endoscopic Scissors Cutting Endoscopic Nasobiliary Drainage Tube in the Treatment of Malignant Hilar Biliary Strictures: a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Application of Endoscopic Scissors Cutting ENBD Tube in the Treatment of Malignant Hilar Biliary Strictures
Acronym: ENBD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit patients
Sponsor: Changhai Hospital (Other)
Collaborators: First People's Hospital of Hangzhou (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Fuzhou General Hospital (Other); LanZhou University (Other); Zhejiang University (Other); Chengdu PLA General Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); General Hospital of Beijing PLA Military Region (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Peking Union Medical College Hospital (Other); ShuGuang Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Xijing Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENBD-01
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; Klatskin Tumor
Keywords: Endoscopic Retrograde Cholangiopancreatography; endoscopic drainage; endoscopic nasobiliary drainage; stent
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic scissors (Experimental): Endoscopic nasobiliary drainage for malignant hilar biliary strictures at first， and application of endoscopic cutting technique followed.
  Interventions: Device: Endoscopic scissors
- Stent (Active Comparator): Standard placement of biliary stent for malignant hilar biliary strictures.
  Interventions: Device: Biliary stent

INTERVENTIONS:
Device: Endoscopic scissors — Application of endoscopic cutting technique following endoscopic nasobiliary drainage in the treatment of malignant hilar biliary strictures.
  Arms: Endoscopic scissors
Device: Biliary stent — Standard placement of biliary stent
  Arms: Stent

SUMMARY:
The purpose of this study is to evaluate application value of the endoscopic cutting technique in the treatment of malignant hilar biliary strictures.

DETAILED DESCRIPTION:
The management unresectable malignant hilar biliary strictures is still very difficult in spite of the rapid development of new endoscopic devices.The application of stent (plastic or metallic) has allowed us to achieve successful drainage. However,there are many complications related to the placement of stents,such as cholangitis,high rate of re-intervention,and so on. The application of endoscopic cutting technique is considered to reduce these complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age over 18 and able to tolerate ERCP.
2. Pathologically confirmed inoperable malignant hilar biliary strictures of Bismuth type II to IV.
3. No history of biliary tract surgery and first attempt at endoscopic or percutaneous drainage.
4. No acute cholangitis before ERCP.
5. Informed consent.

Exclusion Criteria:

1. The patient is very ill(Septic shock, sepsis,coagulation disorders and so on) and cannot tolerate endoscopic treatment.
2. Previous biliary drainage procedure.
3. Inability to provide informed consent.
4. Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
occurrence of acute cholangitis | 30 days
  Acute cholangitis is defined as cholangitis that occurred within 30 days after endoscopic retrograde cholangiopancreatography(ERCP).

SECONDARY OUTCOMES:
Clinical success | 30 days
  Clinical success was defined as a decrease in the total bilirubin level to ≤50% of the pretreatment value within 1 week or to ≤75% within 4 weeks.
Re-intervention | 6 months
  Re-intervention was defined as any type of endoscopic or percutaneous procedure necessary to improve biliary drainage for jaundice or cholangitis after successful placement.

OTHER OUTCOMES:
early adverse | 30 days
  Early adverse event was defined as any ERCP-related adverse event within 4 weeks and a late event was defined as one that occurred after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Department of Gastroenterology, Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uchida N, Ezaki T, Fukuma H, Tsutsui K, Kobara H, Bang MH, Ogawa M, Watanabe K, Ono M, Morishita A, Ogi T, Kamata H, Masaki T, Watanabe S, Kuriyama S. Conversion of endoscopic nasobiliary drainage to internal drainage by means of endoscopic scissor forceps. Endoscopy. 2002 Feb;34(2):180. doi: 10.1055/s-2002-19841. No abstract available. PMID 11822021
- [Background] Kawashima H, Itoh A, Ohno E, Itoh Y, Ebata T, Nagino M, Goto H, Hirooka Y. Preoperative endoscopic nasobiliary drainage in 164 consecutive patients with suspected perihilar cholangiocarcinoma: a retrospective study of efficacy and risk factors related to complications. Ann Surg. 2013 Jan;257(1):121-7. doi: 10.1097/SLA.0b013e318262b2e9. PMID 22895398
- [Background] Asanuma Y, Andoh H, Tanaka J, Koyama K. [Biliary tract cancer]. Nihon Rinsho. 2001 Nov;59 Suppl 7:301-6. No abstract available. Japanese. PMID 11808135